CLINICAL TRIAL: NCT04218006
Title: A Study on the Prevalence of Mutation of Cerebrotendinous Xanthomatosis (CTX) in Families With Kinship Bonds and at Least One Homozygous Patient
Brief Title: A Study on the Prevalence of Mutation of Cerebrotendinous Xanthomatosis (CTX)
Acronym: F-GENE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: TRPHARM (Industry)
Collaborators: Klinar CRO (Other); Damagen Genetic Diagnostic Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: TR-CTX-003
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Xanthomatosis, Cerebrotendinous
Keywords: CTX, Relatives, Index Cases, Kinship, Pedigree
MeSH Terms: conditions — Xanthomatosis, Cerebrotendinous

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specific members of nuclear and extended family relatives will be contacted to propose genetic counseling. Approvals for genetic testing will be asked and necessary information forms will be provided. A total of 5 ml of blood will be collected from each patient for DNA analysis. Blood samples will be analyzed at the Damagen Genetic Diagnosis Center (Ankara), after which no samples will be stored and all samples will be destroyed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Mutation Analysis — Specific members of nuclear and extended family relatives will be contacted to propose genetic counseling. Approvals for genetic testing will be asked and necessary information forms will be provided. A total of 5 ml of blood will be collected from each patient for DNA analysis. Blood samples will be analyzed at the Damagen Genetic Diagnosis Center (Ankara), after which no samples will be stored and all samples will be destroyed.

SUMMARY:
This is a prospective, non-drug epidemological cohort study aimed to investigate the relatives of these cases with CTX-specific gene mutation and clinical features of CTX disease over CTX index cases diagnosed with CTX disease throughout the clinics in Turkey. Relatives included in the study (relatives of CTX index cases) will be taken into clinical and genetic evaluation. Relatives will not receive any experimental intervention or treatment because of their participation in the study. Therefore, this study does not include a treatment protocol or does not have a predetermined visit flow chart. However, relatives of CTX index cases should give consent to genetic testing.

DETAILED DESCRIPTION:
WORK DESIGN STAGES:

1. The CTX index case will be identified and the CTX genetics will be reapproved. The following steps will be provided for all cases.

   * Re-validation of CTX genetics: Cases of CTX indexes that are unrelated and clearly identified the CTX homozygous inheritance identified in the CYP27A1 gene by kinship.
   * Documenting the nuclear and extended family structure and extracting family trees (interview with index cases and parents of index cases)
   * Documentation of all potential symptoms compatible with CTX disease, including data based on the CTX suspicion index (Mignarri Index) in the nuclear and extended family
   * Documentation of patients who have died due to unexpected death or unwillingness to participate in the study.
   * Specific members of nuclear and extended family relatives will be contacted to propose genetic counseling. Approvals for genetic testing will be asked and necessary information forms will be provided. A total of 5 ml of blood will be collected from each patient for DNA analysis. Blood samples will be analyzed at the Damagen Genetic Diagnosis Center (Ankara), after which no samples will be stored and all samples will be destroyed.
   * Collecting blood samples from index cases and, where possible, all nuclear family members (such as parents and siblings)
2. The target cohort will be defined in each family according to the interview results. If the study physician predicts that there are fewer than 50 patients in a large family for the study and follow-up period, this family will be excluded from the study. The initial objective will be to involve grandparents, all their children, married wives and grandchildren. This choice can be adapted by the physician depending on the special situation in the family according to the results of individuals who have undergone genetic mutation tests in the nuclear family, if any, and the definition of nuclear and extended relatives may change in consanguineous families. All extended family members of each identified CTX case will be invited to perform the following steps:

   * Genetic counseling (ideally per family)
   * Approvals for genetic testing will be asked and necessary information forms will be provided. A total of 5 ml of blood will be collected from each patient for DNA analysis. Blood samples will be analyzed at the Damagen Genetic Diagnosis Center (Ankara) and no samples will be stored after the analysis and all samples will be destroyed. Documentation of key data for each case
   * Confirming that the family tree is correctly identified.
   * Documenting patients who have died due to unexpected death or unwillingness to participate in the study.
   * Perform limited neurological examination for key signs and symptoms and document it according to the CTX suspicion index (Mignarri Index).
3. Testing all samples by DNA sequencing for the identified mutation analysis. According to the results, large family cohort will be extracted. In some families, this number can reach up to 600-800 cases.
4. Re-inviting all study cases with disease genotypes for extended neurological examination and medical / genetic counseling.
5. To offer genetic counseling to all study patients with carrier genotypes so that they can make informed decisions about marriage and the next generation (the study coordinator will propose the medical follow-up of new cases diagnosed genetically as CTX).

ELIGIBILITY:
Inclusion Criteria:

* The family of each CTX index case should have more than 50 members in at least three generations.
* CTX index cases should be from different families.
* Index cases and relatives and / or legal representatives are required to be willing to give written informed consent.

Exclusion Criteria:

* Relatives of unconfirmed CTX index cases or non-homozygous CTX patients for disease-causing CTX mutation.
* The patient and / or his / her legal representative does not consent to participate in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The family of each CTX index case should have more than 50 members in at least three generations. All the family members of the CTX index cases will be asked for sampling.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Frequency of CTX mutation | 1 year
  Frequency of CTX mutation (affected or carrier mutation) among relatives

SECONDARY OUTCOMES:
Signs or symptoms compatible with CTX disease | 1 year
  Proportion of cases and relatives with current and / or past signs or symptoms compatible with CTX disease
Mignarri Index | 1 Year
  CTX disease scoring index values
Pedigree | 1 year
  A family tree of the index case

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Onal, Asc. Prof., Principal Investigator — Kanuni Sultan Suleyman University Hospital, Pedaitric Metabolism
Locations (1):
- Osmaniye / Index Case 1 Family Village, Osmaniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided